CLINICAL TRIAL: NCT00619502
Title: Immunogenicity and Safety Study of a Booster Dose of DTaP-IPV-Hep B-PRP~T Combined Vaccine at 15 to 18 Months of Age Following a Primary Series at 2, 3 and 4 Months of Age in Healthy Turkish Infants
Brief Title: Study of Immunogenicity and Safety of a Booster Dose of DTaP-IPV-HB-PRP~T Combined Vaccine in Healthy Turkish Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: A3L22
Record Dates: First submitted 2008-02-11; First posted 2008-02-21 (Estimated); Results first posted 2014-04-03 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-04

CONDITIONS: Diphtheria; Polio; Pertussis; Hepatitis B
Keywords: Hepatitis B; Polio; Diphtheria; Pertussis; H.influenzae type b
MeSH Terms: conditions — Diphtheria; Poliomyelitis; Whooping Cough; Hepatitis B | interventions — DTaP-IPV-HB-PRP-T vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DTaP-IPV-Hep B-PRP~T Vaccine Group (Experimental): Participants received a primary series of 3 vaccinations with DTaP-IPV-Hep B-PRP~T, with 1 dose each at 2, 3, and 4 months of age, in Study A3L10; they will receive a booster dose of DTaP-IPV-HepB-PRP~T at 15 to 18 months of age in the present study
  Interventions: Biological: DTaP-IPV-HB-PRP~T vaccine
- Pentaxim™ + Engerix B™ Vaccines Group (Active Comparator): Participants received a primary series of 3 vaccinations with Pentaxim™ and Engerix B™ vaccines, with 1 dose each at 2, 3, and 4 months of age, in Study A3L10; they will receive a booster dose of DTaP-IPV-Hep B-PRP~T at 15 to 18 months of age in the present study.
  Interventions: Biological: DTaP-IPV-HB-PRP~T vaccine

INTERVENTIONS:
Biological: DTaP-IPV-HB-PRP~T vaccine — 0.5 mL, intramuscular (IM)

SUMMARY:
This is a follow-up of Study A3L10 (NCT00315055)

Immunogenicity

* To describe the antibody persistence following a primary series vaccination of either DTaP-IPV-HB-PRP~T or PENTAXIM™ and ENGERIX B®.
* To describe the immunogenicity of a booster dose of DTaP-IPV-HB-PRP~T.

Safety

- To describe the safety profile after a booster dose of DTaP-IPV-HB-PRP~T.

ELIGIBILITY:
Inclusion Criteria:

* Toddler previously included in Study A3L10 who completed the three-dose primary series vaccination of either DTaP-IPV-HB-PRP~T or PENTAXIM™ and ENGERIX B® at 2, 3 and 4 months of age.
* Toddler of 15 to 18 months of age (range: 456 to 578 days of age inclusive).
* Informed Consent Form signed by the parent(s) or other legal representative(s) and an institution official other than an Investigator.
* Able to attend all scheduled visits and to comply with all trial procedures.

Exclusion Criteria:

* Participation in another clinical trial in the 4 weeks preceding the booster vaccination.
* Planned participation in another clinical trial during the present trial period.
* Congenital or acquired immunodeficiency, immunosuppressive therapy such as long-term systemic corticosteroid therapy.
* Systemic hypersensitivity to any of the vaccine components or history of a life-threatening reaction to a vaccine containing the same substances.
* Chronic illness at a stage that could interfere with trial conduct or completion.
* Blood or blood-derived products received in the last 3 months.
* Any vaccination in the 4 weeks preceding the booster vaccination.
* Any vaccination planned until second Visit.
* History of documented pertussis, tetanus, diphtheria, polio, Haemophilus influenzae type b or hepatitis B infection(s) (confirmed either clinically, serologically or microbiologically).
* Previous booster vaccination against pertussis, tetanus, diphtheria, polio or Haemophilus influenzae type b, and hepatitis B infection(s).
* Coagulopathy, thrombocytopenia or a bleeding disorder contraindicating intramuscular vaccination.
* Any vaccine-related serious adverse event that occurred following the three-dose primary series administration of the investigational vaccine or of the reference vaccine in Study A3L10 (NCT00315055).
* Febrile (temperature ≥ 38.0°C) or acute illness on the day of inclusion.
* Known contraindication to further vaccination with a pertussis vaccine, i.e.: Encephalopathy; temperature > 40.0°C within 48 hours following a vaccine injection, not due to another identifiable cause during the primary series; Inconsolable crying that occurred for > 3 hours within 48 hours following vaccine injection during the primary series; Hypotonic hyporesponsive episode within 48 hours following vaccine injection during the primary series; Seizures with or without fever within 3 days following vaccine injection.

Ages: 15 Months to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 254 (Actual)
Dates: Start 2007-12; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (1):
- Ankara, Turkey (Türkiye)

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 14 December 2007 to 07 January 2008 at 1 clinical center in Turkey.
Pre-assignment Details: A total of 254 participants who met all inclusion, but no exclusion criteria were enrolled and vaccinated.
Groups:
- DTaP-IPV-HepB-PRP~T: All participants received a primary series of 3 vaccinations with DTaP-IPV-HepB-PRP~T, with 1 dose each at 2, 3, and 4 months of age, in Study A3L10; they received a booster dose of DTaP-IPV-HepB-PRP~T at 15 to 18 months of age in the present study.
- Pentaxim™ + Engerix B™: All participants received a primary series of 3 vaccinations with Pentaxim™ and Engerix B™ vaccines, with 1 dose each at 2, 3, and 4 months of age, in Study A3L10; they received a booster dose of DTaP-IPV-Hep B-PRP~T at 15 to 18 months of age in the present study.
Period: Overall Study
Arm/Group | DTaP-IPV-HepB-PRP~T | Pentaxim™ + Engerix B™
Started | 130 | 124
Completed | 122 | 114
Not Completed | 8 | 10
Not completed — Lost to Follow-up | 8 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DTaP-IPV-HepB-PRP~T | Pentaxim™ + Engerix B™ | Total
Number analyzed (Participants) | 130 | 124 | 254
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 130 | 124 | 254
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Months] | 17.6 (0.198) | 17.6 (0.279) | 17.6 (0.241)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 54 | 110
  Male | 74 | 70 | 144
Region of Enrollment [Number; unit: Participants]
  Turkey | 130 | 124 | 254

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Pre-booster Antibody Persistence and Booster Response to DTaP-IPV-Hep B-PRP~T After Primary Vaccination With Either DTaP-IPV-Hep B-PRP~T or Pentaxim™ + Engerix B Vaccine™
Description: Antibody titers measured by chemiluminescence detection for Hepatitis B (Hep B); Farr type radioimmunoassay for Haemophilus influenza type b (PRP); toxin neutralization for Diphtheria (D); indirect enzyme-linked immunosorbent assay (ELISA) for Tetanus (T); neutralization assay for Poliovirus types 1, 2, and 3; and ELISA for Pertussis toxoid (PT) and Filamentous hemagglutinin (FHA). Persistence and response: ≥ 10 mIU/mL for anti-Hep B, ≥ 0.15 µg/mL for anti-PRP, ≥ 0.01 IU/mL for anti-D and anti-T, ≥ 8 (1/dil) for anti-Poliovirus; and ≥ 4-fold increase from Day 0 for anti-PT and anti-FHA.
Time Frame: Day 0 before and Day 30 Post-booster vaccination
Population: Antibody titers were assessed in all participants with any immunogenicity data who did not have any protocol violations that might have interfered with primary criteria evaluation.
Measure: Number; unit: Percentage of Participants
Arm/Group | DTaP-IPV-HepB-PRP~T | Pentaxim™ + Engerix B™
Number analyzed (Participants) | 114 | 103
Percentage of Participants
  Anti-Hep B Pre-booster (N = 109, 103) | 81 | 99
  Anti-Hep B Post-booster (N = 111, 103) | 97 | 100
  Anti-PRP Pre-booster (N = 113,102) | 85 | 83
  Anti-PRP Post-booster (N = 114, 103) | 100 | 100
  Anti-Diphtheria Pre-booster (N = 104, 94) | 90 | 88
  Anti-Diphtheria Post-booster (N = 112, 98) | 100 | 100
  Anti-Tetanus Pre-booster (N = 97, 90) | 100 | 100
  Anti-Tetanus Post-booster (N = 109, 96) | 100 | 100
  Anti-Polio 1 Pre-booster (N = 88, 86) | 99 | 99
  Anti-Polio 1 Post-booster (N = 105, 87) | 100 | 100
  Anti-Polio 2 Pre-booster (N = 84, 87) | 100 | 98
  Anti-Polio 2 Post-booster (N = 101, 83) | 100 | 100
  Anti-Polio 3 Pre-booster (N = 88,86) | 85 | 97
  Anti-Polio 3 Post-booster (N = 102, 84) | 100 | 100
  Anti-PT Post-booster (N = 86, 79) | 97 | 96
  Anti-FHA Post-booster (N = 73,77) | 92 | 97

2. Primary Outcome: Geometric Mean Titers (GMTs) Before and After Booster Vaccination With DTaP-IPV-Hep B-PRP~T
Description: Antibody titers were measured by chemiluminescence detection for Hepatitis B (Hep B); Farr type radioimmunoassay for Haemophilus influenza type b (PRP); toxin neutralization test for Diphtheria (D); indirect enzyme-linked immunosorbent assay (ELISA) for Tetanus (T); neutralization assay for Poliovirus types 1, 2, and 3; and ELISA for Pertussis toxoid (PT) and Filamentous hemagglutinin (FHA).
Time Frame: Day 0 before and Day 30 post-booster vaccination
Population: GMTs were assessed in all participants with any immunogenicity data who did not have any protocol violations that might have interfered with primary criteria evaluation (Per Protocol Population).
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | DTaP-IPV-HepB-PRP~T | Pentaxim™ + Engerix B™
Number analyzed (Participants) | 114 | 103
Titers
  Anti-Hep B Pre-booster (N = 109, 103) | 44.2 [32.3 to 60.7] | 223 [176 to 282]
  Anti-Hep B Post-booster (N = 111, 103) | 1379 [916 to 2078] | 26189 [19133 to 35846]
  Anti-PRP Pre-booster (N = 113, 102) | 0.724 [0.541 to 0.968] | 0.612 [0.443 to 0.844]
  Anti-PRP Post-booster (N = 114, 103) | 72.5 [55.8 to 94.3] | 86.9 [69.8 to 108]
  Anti-Diphtheria Pre-booster (N = 104, 94) | 0.028 [0.022 to 0.035] | 0.032 [0.024 to 0.041]
  Anti-Diphtheria Post-booster (N = 112, 98) | 5.09 [3.89 to 6.66] | 10.2 [7.59 to 13.8]
  Anti-Tetanus Pre-booster (N = 97, 90) | 0.244 [0.204 to 0.292] | 0.194 [0.158 to 0.238]
  Anti-Tetanus Post-booster (N = 109, 96) | 8.98 [7.52 to 10.7] | 13.1 [10.8 to 15.8]
  Anti-Polio 1 Pre-booster (N= 88, 86) | 110 [81.6 to 148] | 114 [82.4 to 157]
  Anti-Polio 1 Post-booster (N = 105, 87) | 5477 [4401 to 6814] | 9050 [7134 to 11480]
  Anti-Polio 2 Pre-booster (N = 84, 87) | 114 [84.9 to 153] | 131 [95.3 to 179]
  Anti-Polio 2 Post-booster (N = 101, 83) | 6099 [4916 to 7566] | 9170 [7170 to 11727]
  Anti-Polio 3 Pre-booster (N = 88, 86) | 47.1 [33.1 to 67.1] | 101 [73.0 to 141]
  Anti-Polio 3 Post-booster (N = 102, 84) | 5542 [4156 to 7392] | 10152 [7806 to 13205]
  Anti-PT Pre-booster (N = 86, 87) | 6.08 [4.74 to 7.79] | 7.49 [5.97 to 9.41]
  Anti-PT Post-booster (N = 113, 95) | 160 [137 to 187] | 237 [202 to 278]
  Anti-FHA Pre-booster (N = 74, 81) | 12.5 [9.59 to 16.4] | 8.18 [6.49 to 10.3]
  Anti-FHA Post-booster (N = 111, 97) | 222 [194 to 254] | 234 [201 to 272]

3. Primary Outcome: Number of Participants With Solicited Injection Site and Systemic Reactions After Booster Vaccination With DTaP-IPV-Hep B-PRP~T
Description: Solicited Injection Site Reactions: Pain, Erythema, Swelling, and Extensive Swelling of Vaccinated Limb. Solicited Systemic Reactions: Pyrexia (Temperature), Vomiting, Crying, Somnolence, Anorexia, and Irritability.
  Grade 3 defined as: Pain, cries when injected limb is moved or movement of limb reduced; Erythema and Swelling, ≥ 5 cm; Extensive Swelling of Vaccinated Limb, All; Pyrexia, ≥ 39ºC; Vomiting, ≥ 6 episodes/24 hours or requiring parenteral hydration; Crying > 3 hours; Somnolence, sleeping most of time or difficult to wake up; Anorexia, refuses ≥ 3 feeds or most feeds; Irritability, inconsolable.
Time Frame: Day 0 up to Day 7 post-booster vaccination
Population: Solicited reactions were assessed in all participants who received a booster dose of DTaP-IPV-Hep B-PRP~T according to the primary series received (Safety Analysis Population).
Measure: Number; unit: Participants
Groups:
- DTaP-IPV-HepB-PRP-T: All participants received a primary series of 3 vaccinations with DTaP-IPV-HepB-PRP~T, with 1 dose each at 2, 3, and 4 months of age, in Study A3L10; they received a booster dose of DTaP-IPV-HepB-PRP-T at 15 to 18 months of age in the present study.
- Pentaxim™ + Engerix B™: All participants received a primary series of 3 vaccinations with Pentaxim™ and Engerix B™ vaccines, with 1 dose each at 2, 3, and 4 months of age, in Study A3L10; they received a booster dose of DTaP-IPV-HepB-PRP-T at 15 to 18 months of age in the present study.
Arm/Group | DTaP-IPV-HepB-PRP-T | Pentaxim™ + Engerix B™
Number analyzed (Participants) | 121 | 111
Participants
  Pain | 56 | 67
  Grade 3 Pain | 4 | 2
  Erythema | 35 | 50
  Grade 3 Erythema | 3 | 4
  Swelling | 26 | 36
  Grade 3 Swelling | 2 | 3
  Extensive Swelling of Vaccinated Limb | 0 | 0
  Pyrexia | 29 | 36
  Grade 3 Pyrexia | 1 | 0
  Vomiting | 13 | 11
  Grade 3 Vomiting | 2 | 2
  Crying | 29 | 35
  Grade 3 Crying | 3 | 4
  Somnolence | 24 | 25
  Grade 3 Somnolence | 2 | 3
  Anorexia | 40 | 43
  Grade 3 Anorexia | 9 | 8
  Irritability | 51 | 61
  Grade 3 Irritability | 5 | 7

ADVERSE EVENTS:
Time Frame: Adverse events data were collected from Day 0 after booster vaccination to up to 6 months after vaccination.
Arm/Group | DTaP-IPV-HepB-PRP~T | Pentaxim™ + Engerix B™
Serious Adverse Events (participants affected / at risk) | 4/130 | 2/124
Other Adverse Events (participants affected / at risk) | 56/130 | 67/124
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DTaP-IPV-HepB-PRP~T (N=130) | Pentaxim™ + Engerix B™ (N=124)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1)
Gastroenteritis rotavirus (Infections and infestations) | 0 (0) | 1 (1)
Poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.00% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DTaP-IPV-HepB-PRP~T (N=130) | Pentaxim™ + Engerix B™ (N=124)
Vomiting (Gastrointestinal disorders) | 13 (13) | 11 (11)
Injection site erythema (General disorders) | 35 (35) | 50 (50)
Injection site pain (General disorders) | 56 (56) | 67 (67)
Injection site swelling (General disorders) | 26 (26) | 36 (36)
Irritability (General disorders) | 51 (51) | 61 (61)
Pyrexia (General disorders) | 29 (29) | 36 (36)
Anorexia (Metabolism and nutrition disorders) | 40 (40) | 43 (43)
Somnolence (Nervous system disorders) | 24 (24) | 25 (25)
Crying (Psychiatric disorders) | 29 (29) | 35 (35)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.